CLINICAL TRIAL: NCT01100125
Title: Comparison Between Sitagliptin Add-on Therapy and Insulin Dose Increase Therapy for Uncontrolled Type 2 Diabetes on Insulin Therapy
Brief Title: Sitagliptin Versus Insulin Dose Increase in Type 2 Diabetes on Insulin Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Assisstant Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH_ENDO2
Record Dates: First submitted 2010-04-05; First posted 2010-04-08 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Diabetes
Keywords: Diabetes; Sitagliptin; insulin; C-peptide
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Sitagliptin Phosphate; Insulin, Long-Acting; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sitagliptin (Experimental)
  Interventions: Drug: sitagliptin
- insulin dose increase (Active Comparator)
  Interventions: Drug: insulin dose increase

INTERVENTIONS:
Drug: sitagliptin — sitagliptin 100mg once daily, orally, for 24 weeks.
  Other Names: Januvia
  Arms: sitagliptin
Drug: insulin dose increase — insulin dose increase
  Other Names: Long acting insulin (Lantus)
  Arms: insulin dose increase

SUMMARY:
It is well established that inhibition of dipeptidyl peptidase (DPP)-IV reduces glucose levels and preserves pancreatic beta cell function in patients with type 2 diabetes. DPP-IV inhibitors stimulate insulin secretion as well as insulin biosynthesis and inhibit glucagon secretion from pancreas by increasing incretin (GLP-1) levels. Recent studies reported that combination therapy with DPP-IV inhibitors and other oral antidiabetic medication have additive or synergistic effects in lowering glycose level, preserving beta-cell mass and function as well as enhancing insulin sensitivity. However, there have been few studies about the glucose lowering effect of DPP-IV inhibitors in patients with type 2 diabetes on insulin treatment.

The researchers hypothesized that DPP-IV inhibitor add-on therapy to insulin treatment may have favorable effects on glucose control and endogenous insulin secretory function in type 2 diabetic patients. The researchers plan to compare between sitagliptin (DPP-IV inhibitor) add-on therapy and insulin dose increase therapy in uncontrolled type 2 diabetes on insulin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1c ≥ 7%
* Age ≥ 18
* Insulin treatment with or without oral antidiabetic medication

Exclusion Criteria:

* Contraindication to sitagliptin
* Pregnant or breast feeding women
* Type 1 diabetes, gestational diabetes, or diabetes with secondary cause
* Chronic hepatitis B or C (except healthy carrier of HBV), liver disease (AST/ALT > 3-fold the upper limit of normal)
* Renal failure (Cr > 2.0)
* Cancer within 5 years
* Not appropriate for oral antidiabetic agent
* Medication which affect glycemic control
* Disease which affect efficacy and safety of drugs
* Other clinical trial within 30 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The change of HbA1C | 24weeks

SECONDARY OUTCOMES:
the number of patients in HbA1C <7% without hypoglycemia | 24 weeks
hypoglycemia(symptoms consistent with hypoglycemia and confirmed by plasma glucose < 72 mg/dL) | 24 weeks
the change of C-peptide | 24 weeks
the change of body weight and waist circumference | 24 weeks
the change of insulin dose | 24 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam

REFERENCES:
- [Derived] Hong ES, Khang AR, Yoon JW, Kang SM, Choi SH, Park KS, Jang HC, Shin H, Walford GA, Lim S. Comparison between sitagliptin as add-on therapy to insulin and insulin dose-increase therapy in uncontrolled Korean type 2 diabetes: CSI study. Diabetes Obes Metab. 2012 Sep;14(9):795-802. doi: 10.1111/j.1463-1326.2012.01600.x. Epub 2012 Apr 18. PMID 22443183